CLINICAL TRIAL: NCT07172178
Title: Anti-PD-1 Antibody Armored γδ T Cells in the Treatment of Malignant Meningioma, a Phase I Clinical Trail
Brief Title: γδ T-PD-1 Ab Cells in the Treatment of Malignant Meningioma
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Fang Liu, MD, Nanjing Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GDT-003-02
Record Dates: First submitted 2025-09-11; First posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Malignant Meningioma
MeSH Terms: conditions — Meningioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- γδ T-PD-1 Ab cells (Experimental): o Cells will be extracted from a healthy donor, followed by ex-vivo expansion, activation and genetic engineering. The ex-vivo expanded γδ T-PD-1 Ab cells will be adoptively transfused to tumor patients.
  Interventions: Biological: γδ T-PD-1 Ab cells

INTERVENTIONS:
Biological: γδ T-PD-1 Ab cells — Patients will receive 6 cycles of ex-vivo expanded γδ T-PD-1 Ab cells treatments,at two-weeks' intervals.γδ T-PD-1 Ab cells are injected through the Ommaya device in a typical 3+3 dose-escalation design(Dose escalation, 1×10^7, 3×10^7, 1×10^8).

SUMMARY:
This study intends to combine the advantages of γδ T cells and PD-1 monoclonal antibody to conduct an exploratory clinical study on the safety and efficacy of PD-1 antibody armored γδ T cells (γδ T-PD-1 Ab cells) in the treatment of malignant meningioma.

DETAILED DESCRIPTION:
This is a single-center, single-arm, phase I clinical trial to evaluate the safety and efficacy of γδ T-PD-1 Ab cells in patients with malignant meningioma. A typical 3+3 dose-escalation design will be used to determine the optimal dose level of γδ T-PD-1 Ab cells based on the incidence of dose-limiting toxicity (DLT). The initial injection dose level will start from 1×10^7 to 1×10^8 in every 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. The patient voluntarily signs the informed consent and can complete the follow-up examination, evaluation and treatment;
2. Age 18-70 years old (both ends included), both male and female;
3. The histopathological diagnosis was malignant solid tumor;
4. Tumor recurrence is confirmed by imaging (MRI) or re-biopsy/surgery;
5. ECOG score 0-2;
6. Expected survival ≥6 months;
7. Have received chemotherapy or targeted therapy more than 4 weeks ago;
8. Organ function requirements:

   Bone marrow function: white blood cell count≥3×109, platelets ≥70×109/L, a hemoglobin (Hb) ≥90g/L; Liver function: total bilirubin ≤1.5 times the upper limit of normal (ULN); Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤3 times ULN; Renal function: serum creatinine level ≤1.5 ULN; Coagulation function: international normalized ratio (INR) does not exceed 1.5 times the upper limit of normal, and activated partial thromboplastin time (APTT) does not exceed 1.5 times the upper limit of normal.

   Cardiac function: left ventricular ejection fraction (LVEF) > 55%
9. Pregnant women of childbearing age must have a negative serum pregnancy test within 28 days before treatment. Any fertile male and female patients must agree to use effective contraceptive methods throughout the study and for at least 12 weeks after the last study administration.

Exclusion Criteria:

1. Intolerance or allergy to any ingredient or similar drug in the treatment plan planned for this study;
2. Major organ dysfunction:

   Cardiac function: Left ventricular ejection fraction (LVEF) ≤ 55%, New York Heart Association (NYHA) grade III or IV congestive heart failure, QTc > 480 msec, other cardiac diseases as determined by the investigator to be unsuitable for inclusion.

   Liver function: Child-Pugh liver function classification C or above. Pulmonary function: Severe respiratory failure affecting other organs.
3. Uncontrolled epilepsy, severe bleeding risk (such as a recent history of cerebral hemorrhage).
4. Active and/or uncontrolled infections (such as tuberculosis, sepsis, opportunistic infections, active hepatitis B virus (HBV) or active hepatitis C virus (HCV) infection, human immunodeficiency virus (HIV) infection, Treponema pallidum (TP) infection).
5. Severe, uncontrolled systemic autoimmune or inflammatory diseases (such as systemic lupus erythematosus, rheumatoid arthritis, ulcerative colitis, Crohn's disease, and temporal arteritis, Guillain-Barré syndrome (GBS), amyotrophic lateral sclerosis (ALS)).
6. Unstable systemic diseases: unstable angina pectoris, cerebrovascular accident or transient ischemia (within 6 months before screening), myocardial infarction (within 6 months before screening), grade III or IV cardiac dysfunction, refractory hypertension (refractory hypertension is defined as: after lifestyle improvement and using appropriate doses of ≥ 4 antihypertensive drugs (including diuretics), blood pressure cannot be effectively controlled after treatment for more than 1 month and still not controlled), severe arrhythmia requiring drug treatment, hepatic arrhythmia, liver disease, kidney disease or metabolic disorders.
7. Patients with other malignant tumors.
8. Major surgeries within 4 weeks before screening that were assessed by the investigator as unsuitable for inclusion.
9. Participated in other interventional clinical studies within 30 days before enrollment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-10-15 (Estimated); Primary Completion 2028-10 (Estimated); Study Completion 2029-10 (Estimated)

PRIMARY OUTCOMES:
Safety evaluation: Incidence of Adverse events (AEs) | 96 weeks
  Therapy-related adverse events will be recorded and assessed according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE, Version 5.0).
Safety evaluation: Dose limited toxicity (DLTs) | 96 weeks
  The incidence, characteristic and severity of DLTs will be recorded and assessed.
Safety evaluation: Maximum-tolerated dose (MTD) | 96 weeks
  MTD or clinical recommended dose will be recorded and evaluated.

SECONDARY OUTCOMES:
Efficacy evaluation: Objective Response Rate(ORR) | 12 weeks
  Objective response rate will be assessed by investigators.
Efficacy evaluation: Disease Control Rate (DCR) | 12 weeks
  Disease Control Rate will be assessed by investigators.
Efficacy evaluation: Progress Free Survival(PFS) | 12 weeks
  Observation for progression-free survival (PFS) will be recorded until 6 months after the start of 1st cycle of treatment.
Efficacy evaluation: Two-year Overall Survival Rate (OS) | 96 weeks
  Observation for overall survival (OS) will be recorded until 24months after the start of 1st cycle of treatment.

IPD SHARING:
Plan to Share IPD: No